CLINICAL TRIAL: NCT01787032
Title: Relative Bioavailability of Single Oral Dose of BI 113608 When Administered Alone or in Combination With Multiple Oral Doses of Ketoconazole or Voriconazole in Healthy Male Subjects (an Open-label, Randomised, Three-period Cross-over Trial)
Brief Title: Drug-drug Interaction Trial of BI 113608 in Combination With Ketoconazole and Voriconazole in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1314.7; 2012-002538-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-01-30; First posted 2013-02-08 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Ketoconazole; Voriconazole

ARMS (3):
- Period 3: BI 113608+Voriconazole (Experimental): tablets with 240 ml water
  Interventions: Drug: BI 113608; Drug: Voriconazole
- Period 2: BI 113608+Ketoconazole (Experimental): tablets with 240 ml water
  Interventions: Drug: BI 113608; Drug: Ketoconazole
- Period 1: BI 113608 (Experimental): tablets with 240 ml water
  Interventions: Drug: BI 113608

INTERVENTIONS:
Drug: BI 113608 — tablet
  Arms: Period 3: BI 113608+Voriconazole
Drug: BI 113608 — tablet
  Arms: Period 2: BI 113608+Ketoconazole
Drug: BI 113608 — tablet
  Arms: Period 1: BI 113608
Drug: Ketoconazole — tablet
  Arms: Period 2: BI 113608+Ketoconazole
Drug: Voriconazole — tablet
  Arms: Period 3: BI 113608+Voriconazole

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of a single oral dose of BI 113608 without and with ketoconazole and voriconazole at steady state. The assessment of safety and tolerability of BI 113608 administered alone and upon co-administration will be an additional objective of this trial.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The primary objective of this trial was to investigate the relative bioavailability of BI 113608 as a single treatment (BI; Treatment A; Reference (R)) and in combination with Ketoconazole (K) (BI + K; Treatment B; Test1(T1)) or Voriconazole (V) (BI + V; Treatment C; Test2 (T2)).
Groups:
- BI 113608/BI 113608 + Ketoconazole/BI 113608 + Voriconazole: The subjects received BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water followed by Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) followed by Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours.
  A wash-out period of at least 6 days was respected between the administrations of BI 113608.
- BI 113608/BI 113608 + Voriconazole/ BI 113608 + Ketoconazole: The subjects received BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water followed by Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) followed by Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours.
  A wash-out period of at least 6 days was respected between the administrations of BI 113608.
- BI 113608 + Ketoconazole/ BI 113608/ BI 113608 + Voriconazole: The subjects received Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours followed by BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water followed by Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours.
  A wash-out period of at least 6 days was respected between the administrations of BI 113608.
- BI 113608 + Ketoconazole/ BI 113608 + Voriconazole/ BI 113608: The subjects received Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) followed by Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours followed by BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water.
  A wash-out period of at least 6 days was respected between the administrations of BI 113608.
- BI 113608 + Voriconazole/ BI 113608/ BI 113608 + Ketoconazole: The subjects received Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours followed by BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water followed by Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours.
  A wash-out period of at least 6 days was respected between the administrations of BI 113608.
- BI 113608 + Voriconazole/ BI 113608 + Ketoconazole/ BI 113608: The subjects received Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) followed by Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours followed by BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water.
  A wash-out period of at least 6 days was respected between the administrations of BI 113608.
Period: Overall Study
Arm/Group | BI 113608/BI 113608 + Ketoconazole/BI 113608 + Voriconazole | BI 113608/BI 113608 + Voriconazole/ BI 113608 + Ketoconazole | BI 113608 + Ketoconazole/ BI 113608/ BI 113608 + Voriconazole | BI 113608 + Ketoconazole/ BI 113608 + Voriconazole/ BI 113608 | BI 113608 + Voriconazole/ BI 113608/ BI 113608 + Ketoconazole | BI 113608 + Voriconazole/ BI 113608 + Ketoconazole/ BI 113608
Started | 3 | 3 | 3 | 3 | 4 | 4
Received R | 3 | 3 | 3 | 3 | 4 | 3
Received T1 | 3 | 3 | 3 | 3 | 3 | 4
Received T2 | 3 | 3 | 3 | 3 | 4 | 4
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The 'treated set' (full analysis set population in the sense of ICH-E9) included all subjects who received at least one dose of trial drug; the safety analysis was based on the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 113608/BI 113608 + Ketoconazole/BI 113608 + Voriconazole | BI 113608/BI 113608 + Voriconazole/ BI 113608 + Ketoconazole | BI 113608 + Ketoconazole/ BI 113608/ BI 113608 + Voriconazole | BI 113608 + Ketoconazole/ BI 113608 + Voriconazole/ BI 113608 | BI 113608 + Voriconazole/ BI 113608/ BI 113608 + Ketoconazole | BI 113608 + Voriconazole/ BI 113608 + Ketoconazole/ BI 113608 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (1.7) | 33.3 (12.3) | 35.0 (6.2) | 35.3 (8.4) | 32.8 (9.9) | 37.3 (12.5) | 36.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 4 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 113608 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: This outcome measure presents the area under the concentration-time curve of BI 113608 in plasma over the time interval from 0 to the last quantifiable data point.
  The parameter dispersion type (standard deviation) is actually intra individual geometric coefficient of variation (intraindividual gCV).
  Statistical analysis 1: The ratio (Other) is calculated as BI+K (T1): BI (R) [%]. Statistical analysis 2: The ratio (Other) is calculated as BI + V (T2): BI (R) [%].
Time Frame: 1 hour before drug administration and 0:25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 and 72 hours after drug administration.
Population: Pharmacokinetic Set (PKS): The 'PK set' included all subjects of the treated set who provided at least one evaluable observation for at least one primary PK endpoint in at least one treatment period without important protocol violations relevant to the evaluation of PK; PK analyses were based on the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hours/litre (nmol*h/L)
Groups:
- BI 113608: The subjects received BI 113608 film-coated tablet 25 mg orally for 1 day (Day 1) orally with 240 mL of water.
- BI 113608 + Ketoconazole: The subjects received Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours.
- BI 113608 + Voriconazole: The subjects received Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) plus BI 113608 (25 mg single dose) for 1 day (Day 1) orally with 240 mL of water after an overnight fast of at least 10 hours.
Arm/Group | BI 113608 | BI 113608 + Ketoconazole | BI 113608 + Voriconazole
Number analyzed (Participants) | 18 | 18 | 18
nanomol*hours/litre (nmol*h/L) | 494 (36.7) | 1840 (36.9) | 1320 (51.4)
Statistical Analysis 1: Comparison: BI 113608 vs BI 113608 + Ketoconazole; Test type: Superiority or Other; ANOVA; A bioequivalence acceptance range was not specified and no hypothesis was tested as the main focus was on estimation; Ratio = 373.66, 90% CI 2-sided [346.029 to 403.507], Standard Deviation 13.2 — ANOVA model on the logarithmic scale: included effects accounting for following sources of variation: 'sequence', 'patients within sequence', 'period' and 'treatment'. Random effect: 'patients within sequences', others considered as fixed effects
Statistical Analysis 2: Comparison: BI 113608 vs BI 113608 + Voriconazole; Test type: Superiority or Other; ANOVA; A bioequivalence acceptance range was not specified and no hypothesis was tested as the main focus was on estimation; Ratio = 266.94, 90% CI 2-sided [243.267 to 292.914], Standard Deviation 16.0 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Maximum Measured Concentration of BI 113608 in Plasma (Cmax)
Description: This outcome measure presents the maximum measured concentration of BI 113608 in plasma.
  The parameter dispersion type (standard deviation) is actually intra individual geometric coefficient of variation (intraindividual gCV).
  Statistical analysis 1: The ratio (Other) is calculated as BI + K (T1): BI (R) [%]. Statistical analysis 2: The ratio (Other) is calculated as BI + V (T2): BI (R) [%].
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/litre (nmol/L)
Arm/Group | BI 113608 | BI 113608 + Ketoconazole | BI 113608 + Voriconazole
Number analyzed (Participants) | 18 | 18 | 18
nanomol/litre (nmol/L) | 102 (55.5) | 267 (41.9) | 218 (54)
Statistical Analysis 1: Comparison: BI 113608 vs BI 113608 + Ketoconazole; Test type: Superiority or Other; ANOVA; A bioequivalence acceptance range was not specified and no hypothesis was tested as the main focus was on estimation; Ratio = 261.34, 90% CI 2-sided [211.692 to 322.633], Standard Deviation 37.3 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 113608 vs BI 113608 + Voriconazole; Test type: Superiority or Other; ANOVA; A bioequivalence acceptance range was not specified and no hypothesis was tested as the main focus was on estimation; Ratio = 213.39, 90% CI 2-sided [175.783 to 259.051], Standard Deviation 34.1 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 113608 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: This outcome measure presents area under the concentration-time curve of BI 113608 in plasma over the time interval from 0 to infinity.
  The parameter dispersion type (standard deviation) is actually intra individual geometric coefficient of variation (intraindividual gCV).
  Statistical analysis 1: The ratio (Other) is calculated as BI + K (T1): BI (R) [%]. Statistical analysis 2: The ratio (Other) is calculated as BI + V (T2): BI (R) [%].
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hours/litre (nmol*h/L)
Arm/Group | BI 113608 | BI 113608 + Ketoconazole | BI 113608 + Voriconazole
Number analyzed (Participants) | 18 | 18 | 18
nanomol*hours/litre (nmol*h/L) | 496 (36.7) | 1850 (36.9) | 1320 (51.4)
Statistical Analysis 1: Comparison: BI 113608 vs BI 113608 + Ketoconazole; Test type: Superiority or Other; ANOVA; A bioequivalence acceptance range was not specified and no hypothesis was tested as the main focus was on estimation; Ratio = 372.88, 90% CI 2-sided [345.456 to 402.477], Standard Deviation 13.1 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 113608 vs BI 113608 + Voriconazole; Test type: Superiority or Other; ANOVA; A bioequivalence acceptance range was not specified and no hypothesis was tested as the main focus was on estimation; Ratio = 266.56, 90% CI 2-sided [242.955 to 292.456], Standard Deviation 16.0 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 113608 in Plasma (Tmax)
Description: This outcome measure presents time from dosing to maximum measured concentration of BI 113608 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Arm/Group | BI 113608 | BI 113608 + Ketoconazole | BI 113608 + Voriconazole
Number analyzed (Participants) | 18 | 18 | 18
hours (h) | 1.25 (74.5) | 1.40 (56.9) | 1.43 (63.9)

5. Secondary Outcome: Terminal Half-life of BI 113608 in Plasma (t1/2)
Description: This outcome measure presents terminal half-life of BI 113608 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Arm/Group | BI 113608 | BI 113608 + Ketoconazole | BI 113608 + Voriconazole
Number analyzed (Participants) | 18 | 18 | 18
hours (h) | 11.0 (28.0) | 9.20 (18.3) | 10.6 (18.8)

ADVERSE EVENTS:
Time Frame: 15 days of treatment (including two 6-days-wash-out periods between BI 113608 treatments) followed by up to 12 days until the end of study. After study completion there was 30 days Adverse Event (AE) follow up period. 57 days on total.
Groups:
- Ketoconazole: The subjects received Ketokonazol film-coated tablet (200 mg bid) (Brand name: Ketokonazol Polfarmex 200 mg film tablets) for 4 days (Days -2, -1, 1, and 2) orally with 240 mL of water after an overnight fast of at least 10 hours.
- Voriconazole: The subjects received Voriconazole (400 mg bid) (Brand name: Vfend® 200 mg film tablets) for 1 day on Day -2 (loading dose) Voriconazole (200 mg bid) for 3 days (Days -1, 1, and 2) orally with 240 mL of water after an overnight fast of at least 10 hours.
Arm/Group | BI 113608 | BI 113608 + Ketoconazole | BI 113608 + Voriconazole | Ketoconazole | Voriconazole
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 3/18 | 3/18 | 5/19 | 9/19 | 12/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 113608 (N=18) | BI 113608 + Ketoconazole (N=18) | BI 113608 + Voriconazole (N=19) | Ketoconazole (N=19) | Voriconazole (N=20)
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 11
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 5 | 3
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes